CLINICAL TRIAL: NCT06481371
Title: A Single-centre Randomised Controlled Study of 4-week Zuojin Pills in Combination With Sodium Rabeprazole Enteric-coated Tablets or Mosapride Citrate for the Treatment of Functional Dyspepsia Combined With Depression
Brief Title: Zuojin Wan Combined With Rabeprazole or Mosapride for the Treatment of Functional Dyspepsia Combined With Depression
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Nanjing First Hospital, Nanjing Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: KY20240613-02-KS-01
Record Dates: First submitted 2024-06-25; First posted 2024-07-01 (Actual); Last update posted 2024-07-01 (Actual); Status verified 2024-06

CONDITIONS: Functional Dyspepsia; Depression
MeSH Terms: conditions — Depression | interventions — mosapride

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- rabeprazole sodium enteric-coated tablets or mosapride citrate (Experimental): For epigastric pain syndrome, Rabeprazole sodium enteric-coated tablets were given as 20mg/dose, 2 times/day.
  Postprandial discomfort syndrome was treated with mosapride citrate, 5mg/dose, 3 times/day, orally before meals.
  The treatment lasted for 4 weeks.
  Interventions: Drug: Rabeprazole sodium enteric-coated tablets; Drug: mosapride citrate
- Chinese medicine combination group (Experimental): In the Chinese medicine combination group, 3g of Zuojinwan was added to the western medicine group twice a day for 4 weeks.
  Interventions: Drug: zuojinwan; Drug: Rabeprazole sodium enteric-coated tablets; Drug: mosapride citrate

INTERVENTIONS:
Drug: zuojinwan — In the Chinese medicine combination group, 3g of Zuojinwan was added to the western medicine group twice a day for 4 weeks.
  Other Names: zuojin pills
  Arms: Chinese medicine combination group
Drug: Rabeprazole sodium enteric-coated tablets — For epigastric pain syndrome
Drug: mosapride citrate — Postprandial discomfort syndrome

SUMMARY:
To evaluate the symptom improvement of Zuojinwan combined with rabeprazole or Zuojinwan combined with a mosapride regimen in patients with functional dyspepsia combined with depression (liver-stomach depression-heat type) using rabeprazole or mosapride regimen as a control, and to compare the patients' adherence to the medication and the adverse effects between the two groups.

DETAILED DESCRIPTION:
Functional dyspepsia (FD) is the highest incidence of functional gastrointestinal disorders (FGIDs), of which the prevalence of FD combined with depression is 16.4%~22.8%, FD etiology is complex and diverse, and in the "Functional Gastrointestinal Disease Rome IV Diagnostic Criteria" released in 2016, it is clearly proposed that its nature is "brain-gut interaction disorder". The "Rome IV Diagnostic Criteria for Functional Gastrointestinal Diseases" released in 2016 explicitly proposed that its essence is "brain-gut interaction disorder", and it is due to the bidirectional regulation of the brain-gut axis that the phenomenon of combined depression is common in FD patients induced by "brain-gut interaction disorder", which is prone to clinical underdiagnosis and misdiagnosis, and also to clinical depression. It is easy to cause clinical underdiagnosis and misdiagnosis, and also brings many challenges to drug treatment. It is feasible to use Zuojinwan combined with rabeprazole sodium enteric-coated capsules or Zuojinwan combined with mosapride citrate tablets for the treatment of FD combined with depression. The aim of this study is to compare the efficacy of Zuojinwan combined with rabeprazole sodium enteric-coated capsules or mosapride citrate for the treatment of FD combined with depression with that of rabeprazole sodium enteric-coated capsules or mosapride citrate treatment alone.

ELIGIBILITY:
Inclusion Criteria:

* (1) Aged between 18 and 65 years; (2) Fulfilment of western medical diagnostic criteria for FD; (3) Meeting the diagnostic criteria for mild depression; (4) Comply with the diagnostic criteria of Liver and Stomach Depression and Heat Disorder in Chinese medicine; (5) A score of 7-17 on the 17-item Hamilton Depression Scale (HAMD-17) (7-17 being mild depression); (6) Good compliance and autonomous behaviour; (7) Enrolled patients must have a diagnosis of gastroscopy, and the gastroscopic diagnosis should be no abnormality or chronic gastritis, no obvious erosion can be seen under the microscope, and there is no obvious atrophy, intestinal epithelial metaplasia, or heterogeneous hyperplasia in the pathological examination. It should be based on the results of gastroscopy in a tertiary-level hospital within 6 months.

Exclusion Criteria:

* (1) HP-positive patients; (2) Dyspepsia caused by organic diseases of the digestive system, such as peptic ulcer, reflux oesophagitis, erosive gastritis (grade 2 or above), atrophic gastritis, gastrointestinal tract tumour, gastrointestinal haemorrhage, hepatic, gallbladder and pancreatic diseases, intestinal obstruction, inflammatory bowel disease, and so on; (3) Systemic diseases affecting the dynamics of the digestive tract, such as diabetes mellitus, chronic renal insufficiency, connective tissue disease, neurological lesions, etc; (4) Those with severe primary heart, brain, liver, lung, kidney, blood or serious diseases affecting their survival; (5) Those with depression, suicidal tendencies and mental disorders who cannot cooperate; (6) Pregnant and breastfeeding women, patients with recent birth plans; (7) Taking drugs that have an effect on the results of this study within 2 weeks before participating in this study; (8) Those who are allergic to or have adverse reactions to the drugs in this study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2024-06-30 (Estimated); Primary Completion 2025-02-27 (Estimated); Study Completion 2025-04-30 (Estimated)

PRIMARY OUTCOMES:
Depressionsymptom scale | Pre-treatment and 4 weeks of treatment
  Hamilton Depression Scale is assessed patients' depressive symptoms pre- and post-treatment.
FD symptom scale | Pre-treatment and 4 weeks of treatment
  The overall score method for the main symptoms was used, and the overall symptoms included postprandial fullness and discomfort, early satiety, mid-upper abdominal pain, and burning sensation in the mid-upper abdomen. The degree and frequency of symptoms were observed before and after treatment
Chinese Medicine Symptoms | Pre-treatment and 4 weeks of treatment
  Evaluation of Chinese medicine symptoms before and after treatment using the Chinese Medicine Symptoms Score Scale

SECONDARY OUTCOMES:
Adverse events during treatment | Pre-treatment and 4 weeks of treatment
  Ask patients about the occurrence of adverse events during treatment

CONTACTS AND LOCATIONS:
Overall Officials: wanli liu, Study Director — The First Affiliated Hospital with Nanjing Medical University

IPD SHARING:
Plan to Share IPD: No